CLINICAL TRIAL: NCT01466764
Title: Immunomodulation, IL-1 Inhibition, and Postoperative Incisional Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to inability to demonstrate benefit in this patient population.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Gary Peltz, Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-10312011-8587
Record Dates: First submitted 2011-11-01; First posted 2011-11-08 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Pain; Inflammation
Keywords: biomarkers
MeSH Terms: conditions — Pain; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anakinra (Active Comparator): Two subcutaneous injections of anakinra (IL-1ra) were given, the first one hour prior to surgery and the second 24 hours after surgery.
  Interventions: Drug: Anakinra
- Saline injection (Placebo Comparator): Two subcutaneous injections of normal saline (same volume as the anakinra group injection) were given, the first one hour prior to surgery and the second 24 hours after surgery.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Anakinra — An injection of 100 mg Anakinra was administered 1 hour prior to surgery and again 24 hours following surgery.
  Other Names: Kineret
  Arms: Anakinra
Other: Normal Saline — An injection of normal saline was administered 1 hour prior to surgery and again 24 hours following surgery.
  Other Names: No other name
  Arms: Saline injection

SUMMARY:
The investigators hypothesize that perioperative administration of anakinra will reduce incisional pain by lowering the concentration of inflammatory mediators in surgical wounds. This knowledge is important because it suggests a new, previously unexplored pharmacological target for the control of postoperative incisional pain.

DETAILED DESCRIPTION:
This study will test whether administration of anakinra, an IL-1 receptor antagonist, will decrease pain and improve wound healing in patients undergoing vascular or orthopedic surgical procedures. The investigators will administer two doses of Anakinra via an injection under the skin, one dose one hour before surgery and a second dose on the first postoperative day (24 hours after surgery). The investigators will remove fluid from the surgical incisions using a small plastic catheter placed under skin during surgery and measure the amounts of pain- causing inflammatory mediators. The investigators will also measure the amount of pain the participant is experiencing using questions about pain intensity and by gently touching the incision to determine sensitivity of the incision site.

ELIGIBILITY:
Inclusion Criteria:

-Patients 18 years of age and older presenting to the Stanford Preoperative Evaluation Clinic prior to elective orthopedic surgical procedures or elective vascular surgical procedures not involving the abdominal aorta or carotid arteries.

Exclusion Criteria:

Patients will be excluded from participation if they have one or more of the following conditions:

1. Evidence of active local or systemic infection as demonstrated by fever, leukocytosis (white blood cell count > 11,000/ul), productive cough, new infiltrate on chest x-ray, or purulent drainage from any source
2. End-stage renal disease
3. A history of diabetic neuropathy
4. A malignancy other than basal cell carcinoma of the skin or in situ carcinoma of the cervix within the previous 5 years
5. Leukopenia (white blood cell count < 2,000/ul)
6. Thrombocytopenia (platelet count < 100,000/ul)
7. Abnormal liver function test result (aspartate aminotransferase or alanine aminotransferase level ≥1.5-fold the upper limit of normal)
8. A history or infection with tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus
9. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Lobato, MD, Principal Investigator — Stanford U
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 13 were enrolled and 3 participants withdrew prior to randomization
Period: Overall Study
Arm/Group | Anakinra | Saline Injection
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anakinra | Saline Injection | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Median (Full Range); unit: years] | 71.4 [52 to 79] | 74 [57 to 89] | 73 [52 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Concentration Levels of Inflammatory Mediators IL-1 Receptor Antagonist (IL-1ra) Present in Human Wounds Following Surgery With and Without the Use of Anakinra.
Description: Tissue samples were collected at the surgical wound site at 3 time points during the 1st 72 hours following surgery. Tissue samples from subjects receiving placebo, and subjects receiving anakinra injections pre, and post op were analyzed for IL-1
Time Frame: Up to 72 hours following surgery
Population: IL-1ra measurements were invalid due to cross-reaction with the assay platform.
Arm/Group | Anakinra | Saline Injection
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Analgesic Consumption During the 72 Hours Following Surgery
Description: Analgesic consumption is reported as the count of participants receiving each analgesic type. Comparisons between the placebo and active drug groups were made at the conclusion of the study.
  PCA/IV: Patient controlled Analgesia/ Intravenous
Time Frame: Up to 72 hours following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Saline Injection
Number analyzed (Participants) | 5 | 5
Participants
  PCA/IV - Dilaudid (mg) | 5 | 4
  PCA/IV - Fentanyl (mcg) | 3 | 1
  PCA/IV - Morphine | 4 | 4
  PO - Oxycontin(tab) | 5 | 4
  PO - Percocet(tab) | 1 | 1
  PO - Acetaminophen(tab) | 3 | 2

3. Secondary Outcome: Post-operative Pain Intensity
Description: Pain was measured on Day 1 and day 2 following surgery using a VAS scale at rest and on stimulation with Visual Analog Scale (VAS) of 1-10 (1=no pain and 10=worst pain)
Time Frame: Up to 72 hours following surgery
Population: Participants with available data were analyzed.
Measure: Mean (Full Range); unit: units on a Visual Analog scale
Arm/Group | Anakinra | Saline Injection
Number analyzed (Participants) | 4 | 5
units on a Visual Analog scale
  Pain Intensity at Rest Day One | 2.25 [0 to 3] | 2.8 [0 to 7]
  Pain Intensity on Stimulation Day One: number analyzed (Participants) | 3 | 5
  Pain Intensity on Stimulation Day One | 7 [5 to 10] | 6.4 [3 to 10]
  Pain Intensity at Rest Day Two | 2.25 [0 to 3] | 3.6 [0 to 7]
  Pain Intensity on Stimulation Day Two: number analyzed (Participants) | 3 | 5
  Pain Intensity on Stimulation Day Two | 3.3 [0 to 6] | 6.2 [3 to 8]

4. Secondary Outcome: Count of Participants Experiencing Wound Infection in the Study From Surgery Till the Time of Discharge From the Hospital
Description: Evaluation of the surgical wound for symptoms of wound infection was made every day during hospitalization. Records from the first post-operative clinic visit were also evaluated for evidence of wound infection.
Time Frame: Up to 72 hours following surgery plus 3 weeks follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Saline Injection
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

5. Secondary Outcome: Count of Participants With Venous Thrombosis After Surgery During Hospitalization
Description: Evaluation of the surgical wound for symptoms of venous thrombosis was made every day during hospitalization. Records from the first post-operative clinic visit were also evaluated for evidence of venous thrombosis.
Time Frame: Up to 72 hours following surgery plus 3 weeks follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Saline Injection
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

6. Secondary Outcome: Assess Rates of Wound Dehiscence
Description: Evaluation of the surgical wound for symptoms of wound dehiscence was made every day during hospitalization. Records from the first post-operative clinic visit were also evaluated for evidence of wound dehiscence.
Time Frame: Up to 72 hours following surgery plus 3 weeks follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Saline Injection
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

7. Secondary Outcome: Total Length of Hospital Stay
Description: Total length of hospital stay for patients enrolled in the study.
Time Frame: Up to approximately 5 days maximum (admittance to discharge)
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Anakinra | Saline Injection
Number analyzed (Participants) | 5 | 5
hours | 75.06 (17.37) | 87.76 (13.8)

ADVERSE EVENTS:
Time Frame: Up to 72 hours following surgery plus 3 weeks follow-up
Description: Adverse event collection was limited to incidence of wound infection, wound dehiscence, and venous thrombosis
Arm/Group | Anakinra | Saline Injection
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
The trial terminated early. We did not expect to see an effect in such a small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No